CLINICAL TRIAL: NCT03287271
Title: ROCKIF Trial: Re-sensitization of Carboplatin-resistant Ovarian Cancer With Kinase Inhibition of FAK
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Michael McHale (Other)
Collaborators: Verastem, Inc. (Industry); Nine Girls Ask (Unknown)
Responsible Party: Sponsor-Investigator, Michael McHale, Clinical Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 170517
Record Dates: First submitted 2017-08-27; First posted 2017-09-19 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; cancer; ovary; carboplatin; paclitaxel; VS-6063; primary peritoneal carcinoma; fallopian tube; defactinib
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms | interventions — defactinib; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Defactinib (VS-6063) +Carboplatin/Paclitaxel (Experimental): Defactinib (VS-6063) +Carboplatin/Paclitaxel
  Interventions: Drug: VS-6063; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: VS-6063 — Phase 1:
  * First 3 patient cohort: VS-6063 200 mg PO twice daily
  * IF TOLERATED, Second 3 patient cohort: VS-6063 400 mg PO twice daily,
  Phase 2:
  VS-6063 400 mg PO twice daily of a 28 day cycle until disease progression or unacceptable toxicity.
  Other Names: defactinib
Drug: Paclitaxel — Phase 1:
  * First 3 patient cohort: paclitaxel 80 mg/m2 infused IV continuously over 1 hour on days 1, 8, and 15 of a 28 day cycle.
  * IF TOLERATED, Second 3 patient cohort: paclitaxel 80 mg/m2 infused IV continuously over 1 hour on days 1, 8, and 15 of a 28 day cycle.
  Phase 2:
  Paclitaxel 80 mg/m2 infused continuously over 1 hour on days 1, 8, and 15 of a 28 day cycle until disease progression or unacceptable toxicity.
  Other Names: Taxol
Drug: Carboplatin — Phase 1:
  * First 3 patient cohort: carboplatin (AUC of 5 mg/mL/min) IV infused continuously over 1 hour on day 1 of a 28 day cycle.
  * IF TOLERATED, Second 3 patient cohort: carboplatin (AUC of 5 mg/mL/min) IV infused continuously over 1 hour on day 1 of a 28 day cycle.
  Phase 2: carboplatin (AUC of 5 mg/mL/min) infused continuously over 1 hour on day 1 of a 28 day cycle until disease progression or unacceptable toxicity.
  Other Names: Paraplatin

SUMMARY:
The purpose of the study is to investigate the combination VS-6063, carboplatin, and paclitaxel. in the treatment of patients with ovarian cancer.

DETAILED DESCRIPTION:
The purpose of the study is to investigate the combination VS-6063, carboplatin, and paclitaxel. in the treatment of patients with ovarian cancer. The study will evaluate whether this regimen is safe. The study will also evaluate whether the regimen can reduce the amount of cancerous cells in your body. If you agree, you will be treated with VS-6063 by mouth, as well as carboplatin and paclitaxel infusions. Carboplatin and paclitaxel are approved by the FDA for the treatment of ovarian cancer. VS-6063 is considered experimental because it is not approved by the FDA for the treatment of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent or persistent epithelial ovarian, fallopian tube or primary peritoneal carcinoma, diagnosed within 6 months of completing their most recent platinum-containing chemotherapy.
* Patients with the following histologic cell types are eligible: Serous adenocarcinoma, endometrioid adenocarcinoma, mucinous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, transitional cell carcinoma, malignant Brenner's Tumor, or adenocarcinoma not otherwise specified (N.O.S.)
* Must have had one prior platinum-based chemotherapeutic regimen for management of primary disease containing carboplatin, cisplatin, or another organoplatinum compound. This initial treatment may have included intraperitoneal therapy, high-dose therapy, consolidation, noncytotoxic agents or extended therapy administered after surgical or non-surgical assessment.
* Must have NOT received more than two total prior lines of cytotoxic chemotherapy for management of recurrent or persistent disease, including retreatment with initial chemotherapy regimens.
* May have received one additional non-cytotoxic regimen for management of recurrent or persistent disease according to the following definition: Non-cytotoxic (biologic or cytostatic) agents include (but are not limited to) hormones, monoclonal antibodies, cytokines, and small molecule inhibitors of signal transduction.
* Women of childbearing potential must have a negative serum pregnancy test prior to study entry and be practicing an effective form of contraception.

Must have adequate:

* Bone marrow function
* Renal function
* Hepatic function
* Neurologic function
* Recovered from effects of recent surgery, radiotherapy, or chemotherapy. All persistent clinically significant toxicities from prior chemotherapy must be less than or equal to Grade 1.
* Free of active infection requiring antibiotics (with the exception of uncomplicated UTI).
* Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration.

Exclusion Criteria:

* Platinum-refractory ovarian, fallopian tube, or primary peritoneal carcinoma.
* Known second primary or prior malignancy diagnosed within 5 years of study start date (other than previously treated non-melanoma skin cancer).
* Current treatment with chemotherapy or radiation therapy. Any prior therapy directed at the malignant tumor, including biologic and immunologic agents, must be discontinued at least three weeks prior to registration.
* History of treatment with known kinase inhibiting agents.
* History of gastrointestinal fistula, hemorrhage, perforation or peptic ulcer disease.
* Patients who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-02-06 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of VS-6063 plus paclitaxel and carboplatin chemotherapy (Measured Via Adverse Events) | 4 years
  Measured Via Adverse Events
Objective response rate (ORR) | 4 years
  ORR by RECIST 1.1.

SECONDARY OUTCOMES:
To assess the toxicity and adverse event profile of VS-6063 plus paclitaxel and carboplatin chemotherapy (Measured Via Adverse Events) | 4 years
  Measured Via Adverse Events
To describe health-related quality-of-life (QoL) outcomes of patients receiving VS-6063 plus paclitaxel and carboplatin chemotherapy. (Measured Via Questionnaire) | 4 years
  Measured Via Questionnaire
progression free survival (PFS) | 4 years
  PFS by RECIST 1.1.
overall survival (OS) | 4 years
  OS by RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Michael McHale, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No